CLINICAL TRIAL: NCT04359901
Title: Sarilumab for Patients With Moderate COVID-19 Disease: A Randomized Controlled Trial With a Play-The-Winner Design
Brief Title: Sarilumab for Patients With Moderate COVID-19 Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Westyn Branch-Elliman (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Westyn Branch-Elliman, Assistant Professor of Medicine, Harvard Medical School; Investigator, VA Boston Center for Healthcare Organization and Implementation Research; Infectious Disease Consultant, VA Boston Healthcare System, VA Boston Healthcare System
Organization: VA Boston Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 3305
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: COVID
MeSH Terms: interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care plus subcutaneous sarilumab (Active Comparator): Standard of care as directed by the treating clinicians, plus sarilumab 400 mg subcutaneous injection. Sarilumab is provided in prefilled syringes/pens containing 200 mg each as is used clinically, and both injections will be given as soon as is convenient after the patient has decided to enroll.
  Interventions: Biological: SARILUMAB
- Standard of care (No Intervention): Standard of care as directed by the treating clinicians.

INTERVENTIONS:
Biological: SARILUMAB — Single dose of 400 mg subcutaneous sarilumab
  Other Names: KEVZARA
  Arms: Standard of care plus subcutaneous sarilumab

SUMMARY:
Objectives: To determine whether blockade of IL-6R is beneficial in patients with COVID-19 infection of moderate severity.

Research Design: Randomized, controlled trial. Two-arm trial comparing standard care alone to standard care with addition of sarilumab (anti-IL6R). The trial will use a randomized play-the-winner design, in which randomization becomes weighted toward the arm that was more effective in previous subjects in the trial.

Methodology Hospitalized patients meeting clinical criteria for moderate disease and testing positive for coronavirus infection. Interventions: sarilumab, 400 mg subcutaneous injection. Standard care is not pre-specified, may vary among patients, and may include agents with anti-viral activity, such as remdesivir or hydroxychloroquine, among others. Up to 120 patients, primary outcome intubation or death within 14 days. All data will be extracted remotely from the electronic health record (EHR).

Clinical Implications: The study has potential to establish IL-6R blockade, delivered subcutaneously, as standard of care in reducing progression to critical illness in patients with moderate COVID-19 disease.

DETAILED DESCRIPTION:
1. Aims/Objectives

   The effectiveness of blockade of IL-6R in treating patients with COVID-19 disease of moderate severity will be tested in a pragmatic and adaptive randomized trial. The primary outcome is intubation or death within 14 days of enrollment OR administration of a rescue dose of IL-6 inhibition if the patient is do-not-resuscitate (DNR)/do-not-intubate (DNI) and the primary team determines it is appropriate based on clinical deterioration. Secondary outcomes include time to hospital discharge if alive, time to clinical recovery as was defined in a recent study, ICU length of stay, time to return to normal or baseline oxygen saturation, and changes in laboratory biomarkers.
2. Background Information

   SARS-COV-2 is a novel human pathogen that emerged at the end of 2019 and rapidly spread worldwide. Clinical disease caused by this novel infection has a high mortality rate, particularly in older adults and in patients with underlying cardiopulmonary disease, populations that are highly prevalent within the VA healthcare system. This creates an urgent need for the VA to quickly and efficiently identify effective therapies to reduce mortality and spread of the disease. Based on in vitro and in vivo data, potential treatment options include anti-viral drugs (such as antimalarials or medications originally developed to treat HIV infection (e.g., lopinavir/ritonavir, remdesivir)), anti-inflammatory drugs, including IL-6 inhibition, and innovations in supportive care, such as placing patients in prone positioning while awake and not intubated. Importantly, in the context of the global pandemic and exponential spread of the disease, clinical trials must be designed in a manner that 1) optimizes outcomes for Veterans, and 2) produces rapid answers, so that effective treatments can be deployed quickly to reduce unnecessary deaths. Based on a review of 384 ongoing clinical trials by the Centre for Evidence-Based Medicine, and a daily search of open clinical trials, many conventional controlled clinical trials of antiviral drugs and cytokine-blocking drugs are in progress and are likely to be completed within a few months; however, it is possible that these trials, which may take months to implement and report results, will not yield any information about how to treat patients until after the peak of the pandemic is over. A secondary challenge is that it is important to identify what works and what does not work quickly, so that manufacturers can understand what medications need to be produced so that supply chains are adequate for treating all patients who might benefit from an intervention. Thus, innovative clinical trial methodologies are needed in order to produce answers in a highly compressed time frame to inform medical decision-making and supply chain management.

   This novel and innovative proposal concerns use and comparison an existing drug (sarilumab) that blocks the receptor for the inflammatory cytokine IL-6. Most studies of IL-6 pathway blockade are using IV medications and include restrictive eligibility criteria and are directed towards patients with severe disease. The investigators hypothesize that patients earlier in the disease course - prior to severe respiratory decompensation - might benefit the most from IL-6 inhibition, and thus are the population included in this pragmatic trial. This study will expand our knowledge and understanding about how IL-6 inhibition can be used to prevent disease progression in patients with moderate disease. It will use a more readily available subcutaneous, longer-acting formulation directed towards patients with moderate disease, of whom 25-35% can progress to severe disease, often rapidly. Eligibility criteria allow for a broad range of underlying choices of other medications, including antiviral medications such as remdesivir and hydroxychloroquine, among others, baseline laboratory values, and comorbidities, reflecting likely real-world clinical use. Thus, this pragmatic project would fill a major gap in research about the clinical care of patients with COVID-19.

   Release of preliminary results to the popular press already necessitated revision of this protocol after only 9 subjects had been enrolled. Interim analysis of a study of sarilumab by its manufacturer has led to revision of the study population and treatment arms. Originally, two doses (200 mg and 400 mg) were tested, and patients with either severe (oxygen requirement and other poor prognostic features) or critical (mechanical ventilation) disease were included. Interim analysis indicated benefit only with 400 mg in critical disease, so that will be the design of the remainder of that trial. In contrast, a study of of a relatively high dose of tocilizumab (8 mg/kg) was reported to be beneficial in a controlled trial of patients varying in severity from critical illness to merely requiring supplementary oxygen. In response, the current study has been modified to allow routine escalation of dosing among a broad range of "moderate" severity short of critical illness. For patients who are critically ill, it is expected that off-label use of a wide range of "heroic" therapies will be tried, including but not limited to cytokine blocking therapies, so exclusion of such patients from this trial does not limit the therapeutic options for such patients, and from a research perspective, such patients have become the focus of the largest ongoing study of sarilumab.
3. Rationale and Purpose

   Severe COVID-19 disease is characterized by a severe acute respiratory distress syndrome (ARDS) followed by a severe cardiomyopathy in many cases. Based on currently available data, it is unclear how much of the respiratory damage in COVID-19 is due to direct effects of SARS-COV-2, or if the primary driver of severe disease is the inflammatory response generated in response to the virus. The key role of inflammation in the progression of the disease is highlighted by recent studies, which demonstrate that patients who progress to requiring ICU-level care no longer have detectable virus present in their respiratory tract. Thus, identifying drugs that could dampen the inflammatory response prior to severe clinical decompensation without adversely affecting clearance of virus would be clinically useful and lead to improved outcomes. Elevated biomarkers of severe inflammation (such as IL-6, CRP, ferritin, and lymphopenia) have been strongly associated with severe disease and increased mortality in patients with COVID-19, and early development of a strong IgG response may paradoxically be a poor prognostic sign during the acute phase of the disease. In contrast, viral load in upper respiratory secretions at baseline is only modestly associated with clinical outcomes, and viral load declines in most patients after presentation, independent of the clinical course of the disease. Severe disease typically arises more than 2 weeks after symptom onset, a time at which virus is usually no longer detectable. These findings suggest that progression to severe disease may be driven more by the inflammatory response to the disease than a direct viral effect, and point to anti-inflammatory drugs as potentially critical therapeutic options. Importantly, high dose glucocorticoids have been found to be ineffective in severe COVID-19 and are associated with somewhat worse outcomes, so other more targeted anti-inflammatory options are urgently needed.

   Blockade of IL-6 signaling is a particularly attractive approach. Sarilumab and tocilizumab are antibodies to the IL-6 receptor (IL-6R), FDA-approved for long-term treatment of rheumatoid arthritis. Tocilizumab has been used open-label with enough anecdotal success in enough patients in China that the manufacturers of sarilumab and tocilizumab have rapidly opened clinical trials in multiple countries at assess efficacy in patients with severe COVID-19 disease. Tocilizumab has also demonstrated efficacy in reducing mortality associated with the cytokine release syndrome in patients receiving CAR-T treatment for cancer, in which the pathogenic pathway is widespread T-cell activation, which leads to production of pleiotropic inflammatory cytokines such as IL-6 by monocytes. Although trials attempting to rescue patients with severe COVID-19 with ARDS and/or cardiomyopathy are essential and are in progress, the ideal population for clinical use may be patients who are not yet critically ill but are at high risk of clinical deterioration due to secondary inflammation.
4. Relevance to Veterans Health

   COVID-19 has a high mortality rate of 2-3% among symptomatic patients. It is expected to have a particularly high mortality in Veterans, because age >60, underlying cardiovascular or lung disease, and obesity are significant risk factors for mortality and clinical deterioration. Thus, advances in care of patients sick enough to be hospitalized yet prior to intubation are expected to have particular benefit for Veterans.
5. Study Design

Design. Prospective, randomized, unblinded interventional clinical trial.

Two arms: standard care, based on established practices within the medical center, or standard care plus subcutaneous sarilumab.

Assignment Strategy: Randomized play-the-winner design, such that randomization becomes weighted toward the arm that was more effective in previous enrolled subjects. The probability of randomization to a specific arm (standard of care or standard of care plus intervention) will be updated based on outcomes in blocks of 10-20 subjects (see Planned Statistical Analyses). The protocol does not include administration of sarilumab or tocilizumab as a "rescue" medication if a patient randomized to standard of care alone deteriorates to the point that the primary outcome (intubation) is met, or if the patient is DNR/DNI and the patient's primary clinical team determines intubation would be performed if the patient's goals of care included intubation. Such patients may receive any treatment per the judgment of their treating physician, and such treatment might include sarilumab or tocilizumab. Use of sarilumab or tocilizumab in this setting will simply be regarded as a treatment failure and not as a protocol deviation.

Data will be extracted remotely from the EHR. No data will be generated specifically for study purposes.

ELIGIBILITY:
Study subjects will be inpatients with confirmed SARS-CoV-2 testing. Testing is performed at the discretion of the treating physician. Only Veterans will be enrolled.

Inclusion Criteria:

1. Positive testing for novel coronavirus SARS-CoV-2019
2. Patients with moderate COVID-19 disease as defined clinically:

   1. Score of 1-3 (out of 3) on a modified Brescia COVID respiratory severity score (BCRSS), elements of which include wheezing or inability to speak complete sentences without effort, respiratory rate ≥22, O2 saturation ≤ 94% with or without supplemental oxygen, or requiring ≥2L supplemental oxygen to maintain O2 Sat >94% in patients without previously documented hypoxia or baseline oxygenation requirement; either is equal to one point on the score) all within a 24-hour period prior to enrollment, and/or any worsening of chest X-ray (CXR) findings after COVID-19 diagnosis
   2. Worsening of baseline oxygenation by at least 3%, or increase in oxygen requirement by at least 2L, in patients with pre-existing hypoxemia or receiving supplemental oxygen chronically.
   3. The BCRSS risk calculation score is available at: https://www.mdcalc.com/brescia-covid-respiratory-severity-scale-bcrss-algorithm

Exclusion Criteria:

1. Critical disease, defined by need for mechanical ventilation
2. Expected death within 48 hours
3. Patients taking any of the following for chronic inflammatory diseases: glucocorticoids equivalent to prednisone > 10 mg/day (methylprednisolone > 8 mg/day, dexamethasone > 2 mg/day), a JAK inhibitor (tofacitinib, baricitinib, upadacitinib), or a biologic

   1. Use of chronic inhaled steroids is NOT an exclusion
   2. Current or recent short-term use of glucocorticoids for chronic conditions such as COPD or gout is NOT an exclusion.
   3. Current use of glucocorticoids for COVID-19 is NOT an exclusion
   4. Use of biologics for non-inflammatory diseases is NOT an exclusion
4. Receipt of any IL-6 inhibitor within 3 months prior to enrollment in the trial
5. Pregnancy, due to lack of fetal monitoring capabilities
6. Patients enrolled in other interventional clinical trials, including for COVID-19. Patients enrolled in non-interventional studies or receiving non-FDA-approved drugs for compassionate use are not excluded.
7. Patients whose goal of care is comfort measures only
8. Inability to provide informed consent, or absence of a legally authorized representative to provide informed consent.
9. Severe psychiatric disease that prevents compliance with typical medical care.
10. Initial positive test for active infection with novel coronavirus SARS-CoV-2019 was >4 weeks prior to current admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Westyn Branch-Elliman, MD, Principal Investigator — VA Boston Healthcare System
Locations (5):
- United States (5):
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - VA Maine Healthcare System, Augusta, Maine
  - VA Boston Healthcare System, Boston, Massachusetts
  - Providence VA Medical Center, Providence, Rhode Island
  - VA Medical Center - White River Junction, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Digital data underlying primary scientific publications will be held as part of a data sharing resource. Study data held for this purpose may include data, data content, format, and organization. The data may contain but are not limited to individually identifiable information, other PHI, and study codes. The data may be available to the public and other VA and non-VA researchers under certain conditions and consistent with the informed consent and CSP policy that prioritize protecting participants' privacy and confidentiality to the fullest extent possible. A detailed plan will be developed in accordance with current technology, infrastructure, best practices, and policies and procedures in place at the time of oversight committee reviews (e.g., Privacy Board, Information Security, and Information Technology standards). The plan will include how data will be discovered, retrieved, analyzed, and managed and will note the materials that are available in machine-readable formats.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of primary publication.
Access Criteria: Consistent with VA Privacy, Regulatory and IT requirements and VHA Handbook 1200.12

REFERENCES:
- [Background] Woods P, Flynn M, Monach P, Visnaw K, Schiller S, Holmberg E, Leatherman S, Ferguson R, Branch-Elliman W. Implementation of documented and written informed consent for clinical trials of communicable diseases: Lessons learned, barriers, solutions, future directions identified during the conduct of a COVID-19 clinical trial. Contemp Clin Trials Commun. 2021 Sep;23:100804. doi: 10.1016/j.conctc.2021.100804. Epub 2021 Jun 26. PMID 34222708
- [Background] Dassum SR, Ferguson R, Woods P, Flynn M, Visnaw K, Holmberg E, Schiller S, Shannon C, Brophy M, Monach P, Leatherman S, Branch-Elliman W; VISN-1 Clinical Trials Network COVID-19 Investigators. Patient- reported reasons for non-participation in a COVID-19 therapeutics clinical trial: Findings from a multi-center investigation. Contemp Clin Trials. 2023 Mar;126:107082. doi: 10.1016/j.cct.2023.107082. Epub 2023 Jan 9. PMID 36632925
- [Background] Dhond R, Acher R, Leatherman S, Page S, Sanford R, Elbers D, Meng F, Ferguson R, Brophy MT, Do NV. Rapid implementation of a modular clinical trial informatics solution for COVID-19 research. Inform Med Unlocked. 2021;27:100788. doi: 10.1016/j.imu.2021.100788. Epub 2021 Nov 12. PMID 34786452
- [Background] Branch-Elliman W, Lehmann LS, Boden WE, Ferguson R, Monach P. Pragmatic, adaptive clinical trials: Is 2020 the dawning of a new age? Contemp Clin Trials Commun. 2020 Jul 17;19:100614. doi: 10.1016/j.conctc.2020.100614. eCollection 2020 Sep. PMID 32724866
- [Background] Branch-Elliman W, Monach PA. Not What Anyone Signed up for: Unnecessary and Insurmountable Barriers Encountered in Conducting Clinical Trials in COVID-19. Narrat Inq Bioeth. 2021;11(1):8-15. doi: 10.1353/nib.2021.0003. No abstract available. PMID 34334456
- [Result] Branch-Elliman W, Ferguson R, Doros G, Woods P, Leatherman S, Strymish J, Datta R, Goswami R, Jankowich MD, Shah NR, Taylor TH, Page ST, Schiller SJ, Shannon C, Hau C, Flynn M, Holmberg E, Visnaw K, Dhond R, Brophy M, Monach PA. Subcutaneous sarilumab for the treatment of hospitalized patients with moderate to severe COVID19 disease: A pragmatic, embedded randomized clinical trial. PLoS One. 2022 Feb 25;17(2):e0263591. doi: 10.1371/journal.pone.0263591. eCollection 2022. PMID 35213547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Plus Subcutaneous Sarilumab | Standard of Care
Started | 20 | 30
Follow up to 14 Days | 15 (Died within 14 days (n=5)) | 28 (Withdrawn (n=1) Died within 14 days (n=1))
Follow up to 30 Days | 14 (Died between 15-30 days (n=1)) | 27 (Died between 15-30 days (n=1))
Completed | 14 | 27
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Plus Subcutaneous Sarilumab | Standard of Care | Total
Number analyzed (Participants) | 20 | 30 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.5) | 70.7 (14.8) | 72.3 (32.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 18 | 28 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 28 | 46
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 17 | 28 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 30 | 50
BMI [Mean (Standard Deviation); unit: kilograms per meter squared] — Body Mass Index in kilograms per meter squared
  kilograms per meter squared | 32.4 (6.4) | 32.9 (6.9) | 32.7 (6.6)
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 3 | 3 | 6
  Former smoker | 11 | 21 | 32
  Never smoker | 6 | 5 | 11
  Unknown | 0 | 1 | 1
Brescia COVID respiratory severity score [Mean (Standard Deviation); unit: units on a scale] — Evaluated within 24-hour period prior to randomization. Range is from 0 (least severe) to 3 (most severe).
  units on a scale | 1.8 (0.6) | 1.7 (0.7) | 1.7 (0.7)
Body temperature [Mean (Standard Deviation); unit: Degrees Fahrenheit] — Determined as closest measurement collected from 24-hours before COVID admission to randomization
  Degrees Fahrenheit | 98.3 (1.3) | 98.3 (1.2) | 98.3 (1.2)
Minimum oxygen saturation on room air [Mean (Standard Deviation); unit: Percent oxygen saturation] — Evaluated within a 24-hour period prior to randomization
  Percent oxygen saturation | 93.4 (2.7) | 93.7 (2.9) | 93.5 (2.8)
Use of oxygen supplementation [Count of Participants; unit: Participants] — Determined as the closest measurement collected from 24-hours before COVID admission to randomization
  Participants | 11 | 15 | 26
Oxygen Concentrator flow rate [Mean (Standard Deviation); unit: L/min] — Determined as the closest measurement collected from 24-hours before COVID admission to randomization
  L/min | 2.7 (1.3) | 2.6 (0.8) | 2.7 (1.1)
Non-invasive ventilatory support [Count of Participants; unit: Participants] — Determined as the closest measurement collected from 24-hours before COVID admission to randomization
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intubation or Death
Description: Composite outcome of number of participants with intubation or death
Time Frame: within 14 Days of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Plus Subcutaneous Sarilumab | Standard of Care
Number analyzed (Participants) | 20 | 30
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Standard of Care Plus Subcutaneous Sarilumab | Standard of Care
All-Cause Mortality (participants affected / at risk) | 6/20 | 2/30
Serious Adverse Events (participants affected / at risk) | 7/20 | 5/30
Other Adverse Events (participants affected / at risk) | 8/20 | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Plus Subcutaneous Sarilumab (N=20) | Standard of Care (N=30)
Oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Worsening of chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Death of unknown cause (General disorders) | 1 (1) | 0 (0)
Respiratory failure, cardiac arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Plus Subcutaneous Sarilumab (N=20) | Standard of Care (N=30)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Defined as neutrophil count <1,000 mcL
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — defined as platelet count <75,000 mcL
Alanine aminotransferase elevation (Hepatobiliary disorders) | 0 (0) | 1 (1) — defined as more than 3-fold of evaluation from baseline value
Non-COVID related infection (Bacterial) (Infections and infestations) | 3 (3) | 5 (6)
Non-COVID related infection (Fungal) (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes virus (Infections and infestations) | 2 (2) | 0 (0)
Hemodialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
ECG abnormality (Cardiac disorders) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT04359901/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04359901/ICF_003.pdf